CLINICAL TRIAL: NCT02359474
Title: Trabectedin Combined With Regional Hyperthermia as Second Line Treatment for Adult Patients With Advanced Soft-tissue Sarcoma
Brief Title: Hyper-Thermia Enhanced Anti-tumor Efficacy of Trabectedin
Acronym: HyperTET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Eric Kampmann, Dr. med., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HyperTET
Record Dates: First submitted 2014-11-10; First posted 2015-02-10 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Sarcoma
Keywords: high-risk soft tissue sarcoma; trabectedin
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin; DNA Breaks, Double-Stranded

ARMS (2):
- Trabectedin with regional hyperthermia (Experimental): Trabectedin 1.5 mg/m², 24 hrs continuous i.v. infusion, repetition after 21 days, until progress of disease.
  Additional treatment with regional hyperthermia (RHT): RHT treatment of the tumor area and the surrounding tissue (41-44°C for 60 min treatment time) is applied at the end of Trabectedin infusion (+/- 4 hrs).
  Interventions: Drug: Trabectedin; Genetic: DNA double-strand breaks
- Trabectedin (Active Comparator): Trabectedin 1.5 mg/m², 24 hrs continuous i.v. infusion, repetition after 21 days, until progress of disease.
  Interventions: Drug: Trabectedin; Genetic: DNA double-strand breaks

INTERVENTIONS:
Drug: Trabectedin
  Other Names: Yondelis
Genetic: DNA double-strand breaks — The rationale for combining Tr and RHT is based on immune mechanisms induced by local heating of which are independent of the anti-tumor effects of Tr. Recent results demonstrate that an acute inflammation at the site of the heated tumor area and "danger signals" are responsible for immune reactions against tumor and metastases (Frey 2012). Abscopal effects after local radiation of tumors with response of distant metastases are induced by similar mechanisms like heat stress (Formenti 2013, Golden 2015). The long-term results for soft-tissue sarcoma are consistent with abscopal effects induced by RHT in a randomized trial compared to chemotherapy alone (Issels 2018).

SUMMARY:
This trial compares trabectedin alone to trabectedin in combination with regional hyperthermia in patients with high-risk soft tissue sarcoma. The study is designed to demonstrate a significant benefit for sarcoma-therapy by adding regional hyperthermia.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically confirmed STS (primary or recurrent), except: Ewing sarcoma, osteosarcoma, skeletal chondrosarcoma (extraskeletal chondrosacomas are included), GIST, dermatofibrosarcoma protuberans, malignant mesothelioma, rhabdomyosarcoma
* Patients after failure of first-line chemotherapy (anthracyclines with/without ifosfamide) with or without RHT
* Progressive or recurrent tumor which is unresectable or only resectable with adverse functional outcome
* After macroscopic incomplete resection or marginal resection (tumor-free margins < 1 cm)
* Prior chemotherapy, including anthracyclines with/without ifosfamide (with or without RHT) or patients who cannot be given these medicines
* At least one tumor manifestation which is eligible for hyperthermia
* Performance status (ECOG) 0,1 or 2
* More than 3 weeks from last treatment
* Neutrophil count ≥ 1,5 G/l, hemoglobin ≥ 9 g/dl, platelets ≥ 100 G/l
* Albumin ≥ 25 g/l, total bilirubin ≤ 1 x ULN, ALT/AST ≤ 2.5 x ULN, AP ≤ 2.5 x ULN, Cockroft and Gault's calculated creatinine clearance ≥ 30 ml/min, CPK ≤ 2.5 x ULN
* Patients with the ability to follow study instructions and likely to attend and complete all required visits
* Written informed consent of the subject

Exclusion Criteria:

* Uncontrolled infection (e.g. active viral hepatitis)
* Unstable cardiac status
* Peripheral neuropathy > grade 2
* Known or persistent abuse of medications, drugs or alcohol
* Other malignancy during the last 5 years (exclusion of basal cell carcinoma or adequately treated cervical carcinoma in situ)
* Prior therapy with Tr or known history of hypersensitivity to drugs with a similar chemical structure
* Pregnancy or breast-feeding
* Females of childbearing potential, who are not using and not willing to use medically reliable methods of contraception for the entire study duration
* Uncontrolled CNS-metastases
* Medical or technical impossibility for hyperthermia to heat the major target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | planned after 46 events after start of recruitment which are expected to occur after 27 month

SECONDARY OUTCOMES:
Radiological response according to RECIST | planned after 46 events after start of recruitment which are expected to occur after 27 month
Overall Survival (OS) | planned after 46 events after start of recruitment which are expected to occur after 27 month
Treatment related toxicity (hematological, renal, hepatic, others) | planned after 46 events after start of recruitment which are expected to occur after 27 month

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Issels, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (5):
- Germany (5):
  - Ludwig-Maximilians University of Munich, Klinikum Großhadern, Munich, Bavaria
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Charité - Universitätsmedizin Berlin, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Universitätsklinikum Erlangen, Erlangen